CLINICAL TRIAL: NCT00995397
Title: Non-inferiority, Monocentric Comparative Open Study of Two Topical Pharmaceutical Preparations (Cream and Lotion) of Dexchlorpheniramine Maleate in the Evaluation of Safety and Efficacy for the Relief of Insect Bite Related-symptoms
Brief Title: Non-inferiority Clinical Trial of Dexchlorpheniramine (Cream Versus Lotion) in the Relief of Insect Bite Related Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Celso Pereira Sustovich, Medical Director, Mantecorp Industria Quimica e Farmaceutica Ltda.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERP 976-08
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Insect Bites
Keywords: Insect bites; Dexchlorpheniramine; Lotion; Cream
MeSH Terms: conditions — Insect Bites and Stings | interventions — dexchlorpheniramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexchlorpheniramine 1% lotion (Experimental)
  Interventions: Drug: Dexchlorpheniramine 1% lotion
- Dexchlorpheniramine 1% cream (Active Comparator)
  Interventions: Drug: Dexchlorpheniramine 1% cream

INTERVENTIONS:
Drug: Dexchlorpheniramine 1% lotion — Small amount applied over the lesion twice a day for 7 days.
  Arms: Dexchlorpheniramine 1% lotion
Drug: Dexchlorpheniramine 1% cream — Small amount applied over the lesion twice a day for 7 days.
  Arms: Dexchlorpheniramine 1% cream

SUMMARY:
Insect bite related symptoms (pruritus and papules) are caused by the release of histamine by mast cells in the skin. Topical anti-histaminics can be used to promote relief of these symptoms. Dexchlorpheniramine maleate 1% cream is a topical anti-histaminic formulation approved by ANVISA in Brazil for the relief of skin irritation and allergies, including the ones caused by insect bites. The aim of the present study is to demonstrate non-inferiority of a new pharmacological preparation of dexchlorpheniramine maleate (1% lotion) with the standard preparation (1% cream) for the relief of insect bite related symptoms and to demonstrate the safety of both preparations.

ELIGIBILITY:
Inclusion Criteria:

* Presence of papules resulting from insect bites within the last 72 hours
* Presence of symmetric lesions to compare one side to the other
* Compliance of the subject to the treatment protocol
* Agreement with the terms of the informed consent by the participants or their legal guardians when younger than 18 years old

Exclusion Criteria:

* Pregnancy or risk of pregnancy
* Lactation
* Use of topical or systemic anti-inflammatory, anti-histaminics or immunosuppressive drugs within the last 48 hours prior to the study
* History of atopy or allergic diseases
* History of allergy of any component of the formulations
* Other conditions considered by the investigator as reasonable for non-eligibility

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
Pruritus intensity at insect bite site, evaluated with a 10 point Visual Analogic Scale (VAS) | 7 days

SECONDARY OUTCOMES:
Composite clinical evaluation of erythema, pruritus and papule formation, performed by the investigator using a 4-point scale for each one of the parameters (absent, mild, moderate, intense). This evaluation constitutes the Insect Bite Score. | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele Ltda., Osasco, São Paulo, Brazil